CLINICAL TRIAL: NCT06222294
Title: A Multi-center, Randomized, Single-blind, Parallel Controlled With Active Drug, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Remimazolam Tosilate for Injection for Sedation in the Intensive Care Unit (ICU)
Brief Title: A Study of Remimazolam Tosilate for Sedation in the ICU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR7056-302
Record Dates: First submitted 2023-12-28; First posted 2024-01-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Sedation in the ICU

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Tosilate for Injection (Experimental)
  Interventions: Drug: Remimazolam Tosilate
- Propofol Medium and Long Chain Fat Emulsion Injection (Active Comparator)
  Interventions: Drug: Propofol Medium and Long Chain Fat Emulsion Injection

INTERVENTIONS:
Drug: Remimazolam Tosilate — Loading dose: 0.08mg/kg Maintenance dose: IV remimazolam tosilate, dose range 0-2.0mg/kg/h, increment or decrement of 0.1-0.2mg/kg/h
  Arms: Remimazolam Tosilate for Injection
Drug: Propofol Medium and Long Chain Fat Emulsion Injection — Loading dose: 0.3-0.5mg/kg Maintenance dose: IV Propofol Medium and Long Chain Fat Emulsion Injection, dose range 0.3-4.0mg/kg/h, increment or decrement of 0.3-0.6mg/kg/h
  Arms: Propofol Medium and Long Chain Fat Emulsion Injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Remimazolam Tosilate for Injection for sedation in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients and/or their guardians are able to provide a written informed consent, understand and agree to comply with the study requirements and protocol.
2. Subjects have been treated with endotracheal intubation and mechanical ventilation, and are expected to receive sedation after randomization at least 6 hours. The target sedation level during the period is -2 ≤ RASS ≤ +1.
3. 18 years to 80 years old, male or female.
4. 18 kg/m2 ≤ BMI ≤ 30 kg/m2.

Exclusion Criteria:

1. Deep sedation is required, or continuous sedation is not needed during the study process.
2. Participants (other than in endotracheal intubation) who are expected to require neuro-muscle blockers during sedation.
3. History of epilepsy or status epilepticus.
4. Myasthenia gravis or a history of myasthenia gravis.
5. Severe arrhythmias or heart disease; the circulatory system is unstable.
6. Subjects with a history of severe cardiovascular disease, or cerebrovascular disease, or neurological disease, or mental illness.
7. Subjects with a history of drug abuse.
8. Organ failure before randomization.
9. Abnormal values of the laboratory examination.
10. Allergic to relevant drugs ingredient or component.
11. Pregnant or nursing women.
12. Subjects who has participated in clinical trials of other interventions recently.
13. Other conditions deemed unsuitable to be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Rate of sedation success, sedation success is defined as the percentage of time maintaining target sedation in the entire drug administering time ≥ 70% without rescue sedation. | within 24 hours after administration of research drug

SECONDARY OUTCOMES:
Percentage of time maintaining target sedation in the entire drug administering time. | within 24 hours after administration of research drug
Percentage of subjects receiving rescue sedation | within 24 hours after administration of research drug
The number of additional doses of the research drug | within 24 hours after administration of research drug]
The total dosage of Fentanyl | within 24 hours after administration of research drug
Wake-up time. | within 6 hours after stopping the research drug
Stopping the research drug to extubation time. | within 6 hours after stopping the research drug
Nursing scale score | follow-up period (approx. 5-10 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided